CLINICAL TRIAL: NCT06188325
Title: A Randomized, Three-Period Crossover Study of Single and Repeated Doses for Three Different Strengths of Eliglustat in Healthy Adult, CYP2D6 Extensive and Poor Metabolizers
Brief Title: A Study to Evaluate Pharmacokinetic Parameters of Eliglustat in Healthy Volunteers Who Are CYP2D6 Extensive or Poor Metabolizers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PKM14281; U1111-1294-8432 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Gaucher's Disease
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): CYP2D6 Extensive metabolizers - dose 1, 2 and 3 of eliglustat
  Interventions: Drug: Eliglustat
- Group 2 (Experimental): CYP2D6 Poor metabolizers - dose 1, 2 and 3 of eliglustat
  Interventions: Drug: Eliglustat

INTERVENTIONS:
Drug: Eliglustat — Pharmaceutical form:Capsule-Route of administration:Oral
  Other Names: GZ385660; Cerdelga

SUMMARY:
The primary objective of the study is to evaluate dose proportionality and pharmacokinetics for three different dose levels of eliglustat after single and repeated administration.

DETAILED DESCRIPTION:
Duration of the study for each subject will be between 42 to 79 days, including a screening period up to 28 days, 3 treatment periods of 7 days each period, a washup period of 7-10 days, and an end-of-study visit 8+/-2 days after the last administration.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 30.0 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history, complete physical examination, laboratory parameters, electrocardiograms (ECG)).
* Having given written informed consent prior to undertaking any study-related procedure
* Having given written informed consent prior to undertaking any study-related procedure

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.

The following classes of drugs administered within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception or menopausal hormone replacement therapy:

* Drugs that are strong inducers of CYP3A (eg, rifampin, carbamazepine, phenobarbital,phenytoin, St. John's Wort).
* Drugs that inhibit CYP2D6 or CYP3A (eg, paroxetine, ketoconazole, fluconazole,ranitidine).
* Drugs that are substrates for P-gp (phenytoin, colchicine and dabigatran etexilate) or CYP2D6 (metoprolol, tricyclic antidepressants such as nortriptyline, amitriptyline, or imipramine, and phenothiazines such as perphenazine and chloropromazine).

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameter: Cmax | Multiple timepoints up to Day 35
  Eliglustat after single and repeated doses: Maximum plasma concentration observed (Cmax)
Pharmacokinetic (PK) parameter: tmax | Multiple timepoints up to Day 35
  Eliglustat after single and repeated doses: Time to reach Cmax
Pharmacokinetic (PK) parameter: AUC0-T | Multiple timepoints up to Day 35
  Eliglustat after single and repeated doses: Area under the plasma concentration versus time curve calculated using the trapezoidal method (AUC0-T)
Pharmacokinetic (PK) parameter: AUC | Multiple timepoints up to Day 35
  Eliglustat after single and repeated doses: Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter: AUClast | Multiple timepoints up to Day 35
  Eliglustat after single and repeated doses: Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast
Pharmacokinetic (PK) parameter: tlast | Multiple timepoints up to Day 35
  Eliglustat after single and repeated doses: Time corresponding to the last concentration above the limit of quantification, Clast
Pharmacokinetic (PK) parameter: CL/F | Multiple timepoints up to Day 35
  Eliglustat after single and repeated doses: Eliglustat after repeated dose: CL/F
Pharmacokinetic (PK) parameter: t1/2z | Multiple timepoints up to Day 35
  Eliglustat after single and repeated doses: Terminal half-life associated with the terminal slope (λz)
Pharmacokinetic (PK) parameter: Ctrough | Multiple timepoints up to Day 35
  Eliglustat after single and repeated doses: Plasma concentration observed just before treatment administration during repeated dosing
Number of participants with treatment emergent adverse events, serious adverse events, and adverse event of special interest | Up to Day 42
  Safety was assessed using clinical laboratory evaluations, ECG parameters, and adverse events spontaneously reported by the subject or observed by the Investigator

CONTACTS AND LOCATIONS:
Locations (1):
- M.D.Covance Clinical Research Unit 1341 W, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org